CLINICAL TRIAL: NCT00819676
Title: Analysis of Exhaled Breath by Biosensors in Adults With Asthma: Observational Part of the Study "Effects of add-on Therapy With Oral Montelukast on the Analysis of Exhale Breath by Biosensors in Adults With Asthma
Brief Title: Analysis of Exhaled Breath by Biosensors in Adults With Asthma
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Paolo Montuschi, M.D. Associate Professor of Pharmacology, Catholic University of the Sacred Heart
Other Study IDs: A/220/2007
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- subjects with asthma
  Interventions: Other: analysis of exhaled breath by biosensors; Other: measurement of exhaled nitric oxide
- healthy subjects
  Interventions: Other: analysis of exhaled breath by biosensors; Other: measurement of exhaled nitric oxide

INTERVENTIONS:
Other: analysis of exhaled breath by biosensors
Other: measurement of exhaled nitric oxide

SUMMARY:
The aim of this study is to investigate the pattern of organic volatile compounds (VOCs) in the exhaled breath detected by biosensors in adults with persistent mild asthma. The analysis of VOCs detected by biosensors in asthmatic adults will be compared with that in a control group of healthy subjects and with exhaled nitric oxide (NO).

Identification of breath VOC patterns may be a completely noninvasive new technique for assessing airway inflammation. A device containing a series of nanosensors can be used for breath analysis of VOC patterns through integration with a suitable algorithm for pattern recognition.

Preliminary data indicate that exhaled breath patterns detected by biosensors in healthy subjects are different from those in patients with asthma. In patients with asthma, analysis of exhaled breath using biosensors will be compared with exhaled NO measurement for studying a possible correlation with an independent method for assessing airway inflammation and with spirometry for assessing a possible correlation with lung function.

Measurement of exhaled NO is a well-established, validated, and standardized method for assessing and monitoring of airway inflammation in patients with asthma who are steroid-naive. In patients with asthma, exhaled NO concentrations are correlated with blood eosinophil cell counts and with airway hyperresponsiveness (AHR).

This study could contribute to the identification and development of a completely new non-invasive technique for assessing airway inflammation with important implications for diagnosis and therapeutic monitoring of patients with asthma.

Establishing the effect of anti-inflammatory drugs on breath analysis by biosensors in patients with asthma is relevant for future studies aimed to use this technique in asthma management.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, at least 15 years of age and no more than 70 years.
* Patient has mild persistent asthma (step 2) of the Guidelines for the Diagnosis and Management of Asthma issued by the National Heart, Lung, and Blood Institute of the National Institutes of Health as defined by a history of symptoms at least once a week but less than daily (step 2) (5).
* Current asthma treatment includes short-acting inhaled β-agonist alone as needed.
* Patient fulfils all the following signs and symptoms of asthma:

  * History of symptoms including, but not limited to dyspnea, wheezing, chest tightness, cough, or sputum production for at least 12 months.
  * A forced expiratory volume in one second (FEV1) of at least 80% of the predicted value (pre-bronchodilator) while withholding β-agonist for at least six hours.
  * Patient has a diagnosis of asthma as defined by 1) an increase in FEV1 or PEF of ≥12% (absolute value), 20 to 30 minutes after inhaled β-agonist administration, OR 2) a positive methacholine PC20 (provocative concentration causing a 20% fall in FEV1) of 8 mg/ml or lower which was performed within the previous 12 months, OR 3) a fall in FEV1 of at least 15% after an exercise challenge which was performed within the previous 12 months. β-agonist reversibility and the methacholine and exercise challenge tests may be satisfied within the previous 12 months if there is adequate source documentation.
  * Patients demonstrate symptoms requiring β-agonist use on ≥2 and ≤6 days of the week for the previous two weeks.
* Patient is able to chew a tablet.
* Patient is judged to be in good, stable physical and mental health (except for his/her asthma) based on the medical history, physical examination, and routine laboratory data, and appears able to successfully complete this trial.
* Ability to perform reproducible spirometry.
* Nonsmoker including no use of smokeless tobacco products in the past year.
* Ability of parent to provide informed consent, as evidenced by signing a copy of the consent form approved by the institutional review board of the subject's respective study institution

Exclusion Criteria: none

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: asthma clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
exhaled nitric oxide | baseline

SECONDARY OUTCOMES:
analysis of breath by biosensors | baseline
FEV1 | baseline
FVC | baseline
FEV1/FVC ratio | baseline
FEF25%-75% | baseline
PEF | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Montuschi, M.D., Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Catholic University of the Sacred Heart, Roma, Italy

REFERENCES:
- [Derived] Montuschi P, Santonico M, Mondino C, Pennazza G, Mantini G, Martinelli E, Capuano R, Ciabattoni G, Paolesse R, Di Natale C, Barnes PJ, D'Amico A. Diagnostic performance of an electronic nose, fractional exhaled nitric oxide, and lung function testing in asthma. Chest. 2010 Apr;137(4):790-6. doi: 10.1378/chest.09-1836. Epub 2010 Jan 15. PMID 20081096